CLINICAL TRIAL: NCT05361889
Title: ReAl-life multIceNter Outcomes Registry for Better antithrOmbotic Strategies in Patients With AF (RAINBOW-AF)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220406
Record Dates: First submitted 2022-04-23; First posted 2022-05-05 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Atrial Fibrillation; Anticoagulant Therapy
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anticoagulation therapy is the most important part of the treatment strategy for atrial fibrillation. Previous studies have confirmed that both warfarin and new oral anticoagulants can effectively prevent stroke in patients with atrial fibrillation. However, the current situation of anticoagulation in atrial fibrillation is not optimistic. This project aims to explore the prevalence of inappropriate doses of anticoagulants in my country. , and the influencing factors related to such doses. By analyzing the status quo, characteristics and influencing factors, suggestions and management plans to promote rational use are put forward to provide certain guidance and help for anticoagulation therapy in patients with atrial fibrillation.

DETAILED DESCRIPTION:
The project is carried out in 30 research centers across the country, and the research object is the prescription/medical order data of real-world atrial fibrillation patients (outpatient and inpatient), including clinical diagnosis, drug use, outpatient and emergency and inpatient records, medical records, as well as laboratory tests, Demographic and other aspects of information, a total of 5000 patients were included, and it is expected to be completed within 3 years. The analysis indicators include patient population distribution, comorbid diseases, concomitant drugs, creatinine clearance rate, proportion of various drugs used, CHA2DS2-VASc score and embolism risk, HAS-BLED score, antithrombotic therapy, etc., to evaluate the influencing factors of inappropriate anticoagulation dose, and to explore the macro trend of anticoagulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with incident (initial diagnosis) AF (Atrial Fibrillation) with electrocardiographic documentation or patients with prevalent (existing diagnosis) AF who had initiation or transition to a NOAC
* Anticipated ability to adhere to local regularly scheduled follow-up visits

Exclusion Criteria:

* Atrial flutter only
* Anticipated life expectancy less than 6 months
* Atrial fibrillation caused by reversible factors, such as hyperthyroidism, acute myocardial infarction, acute pulmonary embolism, etc.
* Active bleeding, such as intracranial hemorrhage, gastrointestinal bleeding, etc.
* Patients with deep vein thrombosis, pulmonary embolism, artificial hip/knee replacement and other anticoagulation indications
* Participation in a randomized trial of anticoagulation for AF at the time of enrollment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: AF patients receiving anticoagulants (outpatient or inpatient) in China
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Prevalence of potentially inappropriate NOAC prescriptions | 3 years
  We will adopt an adaptive design to involve for summary of products characteristics, and perform appropriateness assessments of prevalent NOAC strategies based on indications, NOAC selection, or dosages according to reference materials from approved NMPA labeling recommendations for each agent and 2021 European Heart Rhythm Association (EHRA) Practical Guide on the Use of NOACs in AF Patients.
Patient profiles with NOAC prescriptions | 3 years
  Identify the characteristics of participants who were given appropriate NOAC prescriptions and those who did not from various perspectives: demographics, clinical, medical management, prescription information, therapy, regional differences, types of treating physicians, and NOACs availability.
Number of major bleeding events | 3 years
  Major bleeding will be defined according to International Society of Thrombosis and Hemostasis (ISTH) criteria.

SECONDARY OUTCOMES:
Adverse events | 3 years
  Detailed data on management of NOAC-related adverse events will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Shujuan Zhao, Principal Investigator — Henan Provincial People's Hospital

REFERENCES:
- [Derived] Zhao SJ, Chen BY, Hong XJ, Liu YP, Cai HX, Du S, Gu ZC, Ma PZ. Prevalence, risk factors, and prediction of inappropriate use of non-vitamin K antagonist oral anticoagulants in elderly Chinese patients with atrial fibrillation: A study protocol. Front Cardiovasc Med. 2022 Aug 24;9:951695. doi: 10.3389/fcvm.2022.951695. eCollection 2022. PMID 36093129